CLINICAL TRIAL: NCT00358007
Title: Evaluation of Cone Beam Kilovoltage Imaging During Radiation Therapy for Tumors of the Head and Neck
Brief Title: Use of Cone Beam Kilovoltage Imaging in Patients Receiving Radiation Therapy for Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively Terminated by PI
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06U.195; 2006-10 (Other: CCRRC); JT 1153 (Other: JeffTrial Number)
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Neoplasms
Keywords: Kilovoltage Imaging; Cone-beam CT; CBCT; radiation therapy; head and neck neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cone Beam CT (Experimental)
  Interventions: Device: PTV Reduction

INTERVENTIONS:
Device: PTV Reduction — The margin around the area to be treated with radiation is decreased due the image guidance of the cone beam CT

SUMMARY:
To evaluate the use of cone beam computed tomography in treating head and neck to hopefully reduce side effects

DETAILED DESCRIPTION:
The general purpose of this study is to evaluate Kilovoltage (kv) Imaging, specifically the Cone-beam CT (CBCT) scan device, to assess the accuracy of radiation therapy treatment delivery for patients with head and neck neoplasms

ELIGIBILITY:
Inclusion Criteria:

* any patient receiving radiation therapy for a head and neck tumor assigned to the new Elekta Synergy Linare Accelerator

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pramila Rani Anne, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Den RB, Doemer A, Kubicek G, Bednarz G, Galvin JM, Keane WM, Xiao Y, Machtay M. Daily image guidance with cone-beam computed tomography for head-and-neck cancer intensity-modulated radiotherapy: a prospective study. Int J Radiat Oncol Biol Phys. 2010 Apr;76(5):1353-9. doi: 10.1016/j.ijrobp.2009.03.059. Epub 2009 Jun 18. PMID 19540071
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cone Beam CT: Undergo a cone beam CT scan
Period: Overall Study
Arm/Group | Cone Beam CT
Started | 30
Completed | 28
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.19 (12.21)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Average Interfraction Shift of Patients Undergoing Radiotherapy
Description: Determine the magnitude of the systematic error of patient positioning as determined by cone beam CT (CBCT) and the desired placement based on the treatment planning CT scan.
  Every day, prior to radiation treatment, a CBCT will be performed. The CBCT images will be compared to the radiation therapy planning CT image just taken.
Time Frame: Daily prior to radiation
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 28
millimeters
  Medial-lateral dimension | 1.4 (1.4)
  Superoinferior dimension | 1.7 (1.9)
  Anteroposterior dimension | 1.8 (2.1)

2. Primary Outcome: Average Residual Error Motion of Patients Undergoing Radiotherapy
Description: To determine the magnitude of random variance (random error) in radiotherapy treatment of head and neck neoplasms
Time Frame: Daily after each radiotherapy treatment
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cone Beam CT
Number analyzed (Participants) | 28
millimeters
  Medial-lateral dimension | 0.7 (0.8)
  Superoinferior dimension | 0.9 (0.9)
  Anteroposterior dimension | 0.9 (0.9)

ADVERSE EVENTS:
Arm/Group | Cone Beam CT
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 7/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cone Beam CT (N=30)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cone Beam CT (N=30)
Mucositis (General disorders) | 2 (2)
Dehydration (General disorders) | 4 (4)
Fever (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes